CLINICAL TRIAL: NCT02799537
Title: Comparing the Stanford Letter Project Form to Traditional Advance Directives
Acronym: SLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, VJ Periyakoil, Clinical Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 36786
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Advance Directives; Palliative Care
Keywords: supportive care; palliative care; goals of care; advance care planning; advance directives
MeSH Terms: interventions — Advance Directives

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm complete the Stanford letter advance directive
  Interventions: Other: Randomized clinical study
- Control (Active Comparator): Participants in the control arm complete the California state traditional advance directive
  Interventions: Other: Randomized clinical study

INTERVENTIONS:
Other: Randomized clinical study — Participants will be randomly assigned to one of two advance directives and we will assess which they prefer. This is not a human health intervention
  Other Names: Advance Directive

SUMMARY:
Our goal is to compare two types of advance directives forms available in English and Spanish to determine which is more easy to use for patients.

DETAILED DESCRIPTION:
Step1: Any adult participant who is interested in completing advance directives and able to read and write in English and or Spanish will be eligible to participate in the study

Step 2:

Online Stanford consent form will be presented before the participants. Only after they read the consent and click on the participation link will they be able to enter the study.Those who are willing to participate will be randomly assigned to either the letter or traditional advance directives in Spanish and study measures. They will also answer questions as to how much they liked and understood the documents.

Step 4: The investigators will collect data until the investigators reach an n=1000

Step 5: The investigators will analyze the results and submit for publication.

In this protocol, we are assessing whether patients prefer the traditional advance directives or the letter directive. As it is just an questionnaire based study, there no risk for patients.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age

Exclusion Criteria:

* Under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-02; Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Ease of use of Questionnaire. more patient-centered and family oriented | 1year
  It was easy to read and understand the form of advance directive .◦This is a feasibility trail. On completion of the advance directive they were assigned ( letter directive or traditional directive, we are asking questions to participants about whether the directive was clear and easy to understand).

SECONDARY OUTCOMES:
Ease of use to describe how decisions are made | 1year
  Advance form helped me to describe how decisions are made
Ease of use about the type of treatment and care. | 1year
  Advance form stimulated my own thinking about the type of treatment and care they wish to receive in my last days of life.
Ease of use about letting my doctors about my wishes. | 1 year
  This form can help my doctors understand what treatments would like to receive and what not wish to receive in my last days of life ( resuscitation , respirators , artificial feeding , renal dialysis).
Ease of use if I cannot make decisions for myself then the form says it. | 1 year
  In the future, if I can not make decisions for myself, this form will help my family / friends understand exactly what treatments ( resuscitation , respirators , artificial feeding , renal dialysis) would like to receive and what treatments do not wish to receive so they can make decisions medical for me.
Ease of use about my future preferences. | 1 year
  There were issues with my future preferences that were not covered in the form of advance directive .
Ease of use of the form itself. | 1 year
  I feel comfortable using form for advance care planning .
Ease of use and the comments participants may have. | 1 year
  Any comments participants may have about the form of advance directive ? What can investigators do for patients and their families understand it better?

CONTACTS AND LOCATIONS:
Overall Officials: VJ Periyakoil, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This site contains the English and Spanish versions of the letter directive. — http://med.stanford.edu/letter.html
- See also: This site contains the English and Spanish versions of the traditional advance directive. — https://oag.ca.gov/sites/all/files/agweb/pdfs/consumers/ProbateCodeAdvancedHealthCareDirectiveForm-fillable.pdf